CLINICAL TRIAL: NCT05476081
Title: A REAl-life Study on Short-term Dual Antiplatelet Treatment in Patients With Ischemic Stroke or Transient Ischemic Attack
Brief Title: A REAl-life Study on Short-term DAPT in Patients With Ischemic Stroke or TIA
Acronym: READAPT
Status: Completed | Type: Observational
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Simona Sacco, Professor, University of L'Aquila
Other Study IDs: 03/2021
Record Dates: First submitted 2022-07-24; First posted 2022-07-27 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Ischemic Stroke; TIA
Keywords: DAPT; Stroke; TIA; antiplatelet treatment
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Aspirin; Clopidogrel; Ticagrelor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients (single cohort study): Patients presenting with a mild-to-moderate ischemic stroke or high risk TIA
  Interventions: Drug: Aspirin; Drug: Clopidogrel; Drug: Ticagrelor

INTERVENTIONS:
Drug: Aspirin — Aspirin (100-300 mg) administered for 21-90 days in combination with another antiplatelet treatment
  Other Names: B01AC06; acetylsalicylic acid
Drug: Clopidogrel — Clopidogrel (75-600 mg) administered for 21-90 days in combination with another antiplatelet treatment
  Other Names: B01AC04
Drug: Ticagrelor — Ticagrelor (90-180 mg) administered for 21-90 days in combination with another antiplatelet treatment
  Other Names: B01AC24

SUMMARY:
The REAl-life study on short-term Dual Antiplatelet treatment in Patients with ischemic stroke or Transient ischemic attack (READAPT) is an observational, multicenter, prospective study involving Italian centers. The study aims at evaluating effectiveness and safety of short-term (21-90 days) dual antiplatelet treatment (DAPT) in secondary prevention of mild-to-moderate ischemic stroke or high-risk TIA.

DETAILED DESCRIPTION:
The READAPT will depict the benefit/risk profile of DAPT in a clinical setting, and address subgroups of patients such as those with small cerebral vessel diseases or those treated with revascularization procedures.

Randomized clinical trials (RCTs) proved that short-term DAPT is superior over single antiplatelet treatment in reducing the ischemic recurrence risk, without a remarkable increased hemorrhagic risk thanks to the short treatment course. However, RCTs excluded patients treated with revascularization procedures (i.e. intravenous thrombolysis and thrombectomy), did not provide data on neuroimaging, and had slightly different treatment procedures such as time-to-DAPT start and antiplatelets loading dose.

The study comprises a baseline coinciding with the index event, when the investigators will collect demographics and characteristics of the event, and a 90±5 day follow-up from the index event, when patients will be screened for treatment compliance, tolerability and ischemic or hemorrhagic events. Follow-up visit can be performed remotely.

The investigators did not establish strict NIHSS or ABCD2 score cutoff for patients' inclusion, as treatment decision has to be taken independently from the study, and highly recommend physicians to adhere to guidelines. Each participating center will include all consecutive patients (hospitalized or non-hospitalized) who will meet inclusion criteria.

Data were entered in an electronic anonymized database created on the Research Electronic Data Capture (REDCap) software for the analyses hosted at University of L'Aquila. The local PI or the co-investigators will be able to upload patients' data through a single form specifically created for the study, which will include a user-friendly drop-down menu. Anonymized data will be stored on a secured server under the responsibility of University of L'Aquila. The data will be automatically backed-up once a week. Data will not be shared with unauthorized persons. Plausibility of the entered data will be checked by the study manager and the statistical data manger and data queries will be resolved by Local PI. Cases with missing data or unresolved queries will be rejected to retain only the highest quality data in the registry. Data from centers not ensuring consecutive recruitment of patients or adequate follow-up will not be included in the final database.

All analyses will be performed according to the intention-to-treat principle in all included patients completing the 90-day follow-up or having a fatal outcome event within 90 days. Descriptive statistics will be used to report baseline information. The investigators will analyze the time from index event to the first occurrence of primary and secondary outcome events with the use of a Cox proportional hazards model. Two statistical models will be used: Model 1 unadjusted and Model 2 adjusted for demographics and characteristics of the index event. P values for interaction will be calculated according to the following subgroups: type of event (ischemic stroke vs TIA), time to DAPT (≤24 hours vs >24 hours from symptom onset), type of DAPT (aspirin+clopidogrel vs aspirin+ticagrelor), DAPT duration (≤21 vs >21 days and ≤30 vs >30 days), NIHSS score at onset (≤3 vs >3 and ≤5 vs >5), revascularization procedure (i.v. thrombolysis and/or mechanical thrombectomy vs no interventions). Hazard ratios with 95% confidence intervals will be reported. Should multiple events of the same type occur, the time to the first event will be used in the model. Data from patients who had no events during the study will be censored at the time of study termination or death. Assuming a 95% confidence interval, an estimated sample size of 1067 subjects would be required to detect a conservative 50% proportion of primary outcome occurrence with a two-sided 2.5% margin of error.

ELIGIBILITY:
Inclusion Criteria (all to include the patient):

* Patients with mild or moderate non-cardioembolic ischemic stroke or high-risk TIA treated with a short course of DAPT (usually 21-30 days but up to 90-day at the physician's discretion) for the acute event;
* Male or female aged >18 years;
* Providing signed and dated informed consent;
* Willing to comply with all study procedures and to be available for the duration of the study.

Exclusion Criteria (one sufficient to exclude the patient):

* Patients receiving DAPT after endovascular procedures with stenting;
* Patients participating to any interventional RCT on stroke prevention;
* Presence of any condition which may preclude reliability of the collected information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a mild-to-moderate ischemic stroke or high risk TIA (according to the NIHSS Stroke scale and ABCD2 score respectively) receiving 21/90-day DAPT as secondary prevention according to clinical practice. No cutoffs of NIHSS score or ABCD2 score have been established, but we recommend to follow international guidelines.
Sampling Method: Probability Sample
Enrollment: 2239 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Primary composite outcome | 90 days from DAPT start
  Death, stroke recurrence (ischemic or hemorrhagic)

SECONDARY OUTCOMES:
Ischemic stroke | 90 days from DAPT start
TIA | 90 days from DAPT start
Intracerebral hemorrhage (ICH) | 90 days from DAPT start
  Lobar or non lobar ICH
Subarachnoid hemorrhage | 90 days from DAPT start
Other intracranial hemorrhage | 90 days from DAPT start
  Subdural or epidural hematoma
Mild bleeding | 90 days from DAPT start
  bleeding not requiring blood transfusion or causing hemodynamic compromise
Moderate bleeding | 90 days from DAPT start
  bleeding requiring blood transfusion, but not causing hemodynamic compromise
Severe bleeding | 90 days from DAPT start
  bleeding causing hemodynamic compromise and requiring blood transfusion, inotropic support, or surgical intervention and
Myocardial infarction | 90 days from DAPT start
Hospitalization | 90 days from DAPT start
  hospitalization due to any cause
Death due to vascular causes | 90 days from DAPT start
  Death due to stroke (ischemic or hemorrhagic), systemic hemorrhage, myocardial infarction, congestive heart failure, pulmonary embolism, sudden death, or arrhythmia.
Death due to non-vascular causes | 90 days from DAPT start
  Death due all the other causes (i.e. infections, neoplasms etc)

OTHER OUTCOMES:
Modified Rankin Scale (mRs) | 90 days from DAPT start
  measure of the disability through a scale from 1 to 6, where 6 indicated death
Early DAPT discontinuation | 90 days from DAPT start
  Treatment discontinuation due to adverse events, lack of compliance or Diagnosis of atrial fibrillation or other condition requiring anticoagulant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Simona Sacco, MD, Study Chair — Department of Biotechnological and Applied Clinical Sciences, University of L'Aquila
Locations (127):
- Italy (127):
  - Neurology e Stroke Unit Departement, SS Filippo e Nicola Hospital, Avezzano, Abruzzo
  - Department of Neurology and Stroke Unit, Ente Ecclesiastico ospedale Generale Regionale Miulli, Acquaviva delle Fonti
  - Department f Neurology, AO Nazionale SS Biagio and Cesare Arrigo, Alessandria
  - Department of Neurology, Murgia Hospital Fabio Perinei SS 96, Altamura
  - Department of Neurology and Stroke Unit Ospedali Riuniti Ancona, Ancona
  - Department of Neurology, INRCA-IRCCS "U Sestili" Hospital, Ancona
  - Department of Neurology and Stroke Unit, "U. Parini" Hospital, Aosta
  - Department of Neurology, San Donato Hospital, Azienda USL Toscana Sud Est, Arezzo e Val D'Arno, Arezzo
  - Department of Neurology and Stroke Unit, "Di Venere" Hospital, Bari
  - Stroke Unit, Policlinico di Bari, Giovanni XXIII Hospital, Bari
  - Department of Neurology and Stroke Unit, "Mons. Dimiccoli" Hospital, Barletta
  - Department of Neurology,San Bassiano Hospital, Bassano del Grappa
  - Stroke Unit, San Martino di Belluno Hospital ULSS 1, Belluno
  - Department of Neurology, AO San Pio, Benevento
  - Department of Neurology and Stroke Unit, Maggiore Hospital, IRCCS Istituto delle Scienze Neurologiche di Bologna, Bologna
  - Department of Neurology, Policlinico S. Orsola-Malpighi-Clinica Neurologica Metropolitana, IRCCS Istituto delle Scienze Neurologiche di Bologna, Bologna
  - Stroke Center, Gubbio-Gualdo Tadino Hospital, Branca
  - Neuro-vascular Unit, AO Spedali Civili, Brescia
  - Stroke Unit, ASST Franciacorta, Brescia
  - Stroke Unit, Istituto Ospedaliero Fondazione Poliambulanza, Brescia
  - Stroke Unit, A. Perrino Hospital, Brindisi
  - Department of Neurology and Stroke Unit, AO "G. Brotzu", Cagliari
  - Department of Neurology and Stroke Unit, S Elia Hospital, Caltanissetta
  - Stroke Unit, AO San Sebastiano AORN Caserta, Caserta
  - Department of Neurology, San Giacomo Hospital, Castelfranco Veneto
  - Department of Neurology, AO Cannizzaro, Catania
  - Department of Neurology, Institute G. Giglio di Cefalù, Cefalù
  - Department of Neurology and Stroke Unit, "Bufalini" Hospital, Cesena
  - Department of Neurology and Stroke Unit, SS Annunziata Hospital, Chieti
  - Department of Neurology and Stroke Unit, Cittadella, AULSS6 Euganea, Cittadella
  - Stroke Center, USL umbria 1, Città di Castello
  - Stroke Unit, Valduce Hospital, Como
  - Department of Neurology, Conegliano Hospital Aulss 2 Veneto, Conegliano
  - Department of Neurology and Stroke Unit, ASST Maggiore Hospital of Crema, Crema
  - Department of Neurology, ASST Cremona, Cremona
  - Department of Neurology, Santa Croce Hospital, Cuneo
  - Department of Neurology and Stroke Unit, Desio Hospital ASST Monza, Desio
  - Department of Neurology, ASUR Area Vasta 4 (ex ZT11), Fermo
  - Department of NeurologY, AOU of Ferrara, Ferrara
  - Department of Neurology, San Giovanni di Dio Hospital, Florence
  - Stroke Unit, AOU Careggi, Florence
  - Department of Neurology, Ente Ospedali Galliera Genova, Genova
  - Stroke Unit, San Martino Hospital of Genova, Genova
  - Department of Neurology, ASUGI, Gorizia
  - Department of Neurology, USL Toscana sud est, Grosseto
  - Department of Neurology and Stroke Unit, ASUR Marche AV2 Jesi, Iesi
  - Department of Neuology, Sant'Andrea Hospital, Azienda Sanitaria Locale n. 5 "Spezzino" La Spezia, La Spezia
  - Department of Neurology, F Renzetti Hospital, Lanciano
  - UTN, Santa Maria Goretti Hospital, Latina
  - Department of Neurology, Ospedale Vito Fazi, Lecce
  - Department of Neurology, Legnago Hospital, Legnago
  - Department of Neurology and Stroke Unit Ospedale of Legnano, Legnano
  - Emergency Department, Azienda USL 6 Livorno, Livorno
  - Department of Neurology, Valle del Serchio Hospital, Lucca
  - Departement of Neurology, San Salvatore Hospital, L’Aquila
  - Department of Neurology, Apuane Hospital, Azienda USL Toscana Nord Ovest, Massa
  - Department of Neurology, ASST Melegnano e della Martesana, Melegnano
  - Department of Neurology, ASST Merate, Merate
  - Stroke Unit, AOU Gaetano Martino, Messina
  - Stroke Unit, Angelo's Hospital, Mestre
  - Stroke Unit, Istituto Clinico Città Studi, Milan
  - Department of Neurology and Stroke Unit, Humanitas, Milan
  - Department of Neurology and Stroke Unit, IRCCS Istituto Auxologico Italiano, San Luca Hospital, Milan
  - Department of Neurology, Mirano ULSS 3 Serenissima, Mirano
  - Stroke Unit, "S.Agostino-Estense" Hospital, AOU of Modena, Modena
  - Stroke Unit, Santa Croce Hospital, Moncalieri
  - Department of Neurology, San Gerardo Hospital and Bicocca University, Monza
  - Department of Neurology and Stroke Unit, Cardarelli Hospital, Napoli
  - Stroke Unit, Ospedale del Mare, Napoli
  - Department of Neurology and Stroke Unit, AOU Maggiore della Carità, Novara
  - Stroke Unit, San Giacomo Hospital, Novi Ligure
  - Stroke Unit, AOU San Luigi Gonzaga, Orbassano
  - Stroke Unit, Azienda Ospedale Università, Padua
  - Department of Neurology and Stroke Unit, ARNAS Civico of Palermo, Palermo
  - Department of Neurology, Villa Sofia Hospital, Palermo
  - Department of Neurophysiopathology and Stroke Unit, AOUP Paolo Giaccone, Palermo
  - Stroke Unit, Buccheri La Ferla Hospital, Palermo
  - Department of neurology, Azienda Ospedaliero-Universitario di Parma, Parma
  - Stroke Unit, Fidenza AUSL PR, Parma
  - Cerebrovascula disease and Stroke Unit neurological Intitute IRCCS Mondino, Pavia
  - Stroke Unit, AOUUD Santa Maria della Misericordia, Perugia
  - Department of Neurology ande Stroke Unit, Pescara Hospital, Pescara
  - Stroke Unit, Pederzoli Hospital, Peschiera del Garda
  - Department of Neurology, AUSL Piacenza, Piacenza
  - Departement of Neurology and Stroke Center, S.Corona Hospital, Pietra Ligure
  - Department of Neurology and Stroke Unit, E. Agnelli Hospital, Pinerolo
  - Department of Neurology, Azienda ospedaliera e universitaria Pisana, Pisa
  - Department of Neurology, San Jacopo Hospital, Pistoia
  - Stroke Unit, AO"San Carlo", Potenza
  - Department of Neurology, Maria Paternò Arezzo Hospital, Ragusa
  - Department of Neurology and Stroke Unit, Santa Maria delle Croci Hospital, Ravenna
  - Stroke Unit, AO "Bianchi-Melacrino-Morelli", Reggio Calabria
  - Department of Neurology and Stroke Unit, Arcispedale Santa Maria Nuova, Reggio Emilia
  - Department of Neurology, Infermi di Rimini Hospital, Rimini
  - Unità di trattamento neurovascolare, Azienda Ospedaliero Universitaria Policlinico Umberto I, Roma
  - Department of Neurology and Stroke Unit, Sant'Eugenio Hospital, Rome
  - Department of Neurology and Stroke Unit, Systems Medicin, Policlinico Tor Vergata, Rome
  - Department of Neurology, Ospedale Fatebenefratelli, Rome
  - Department of Neurology, Policlinico Gemelli, Rome
  - Department of Neurology, SS Filippo Neri Hospital, Rome
  - Stroke Unit, AO San Camillo, Rome
  - Stroke Unit, AOU Sant'Andrea, Rome
  - Stroke Unit, Ospedale Rovigo, ULSS 18, Rovigo
  - Department of Neurology, Presidio ospedaliero Umberto I Nocera Inferiore, Salerno
  - Department of Neurology, Madonna del Soccorso Hospital, San Benedetto del Tronto
  - Department of Neurology, ASST Lariana, Sant'Anna Hospital, San Fermo della Battaglia
  - Department of Neurology, Casa sollievo della sofferenza, San Giovanni Rotondo
  - Stroke Unit, AOU, Sassari
  - Department of Neurology, SS. Annunziata Hospital, Savigliano
  - Stroke Unit, Azienda ospedaliera universitaria Senese, Siena
  - Department of Neurology, SS Annunziata Hospital, Sulmona
  - Department of Neurology and Stroke Unit, Umberto I Hospital, Syracuse
  - Department of Neurology and Stroke Unit, AO Santa Maria of Terni, Terni
  - Department of Neurology and Stroke Unit, San Giovanni Bosco Hospital, Torino
  - Neuro-vascular Unit, Maria Vittoria Hospital, Torino
  - Department of Neurology and Stroke Unit, ASP of Trapani, Trapani
  - Stroke Unit, Santa Chiara Hospital, Trento
  - Department of Neurology, Cà Foncello Hospital, Treviso
  - Department of Neurology, Azienda Ospedaliera-Universitaria Giuliano Isontina, Trieste
  - Department of Neurology and Rehabilitation, ASUR, Udine
  - Department of Neurology and Stroke Unit, ASST Settelaghi, Varese
  - Department of Neurology, SS Giovanni e Paolo Hospital, Aulss3 Serenissima Veneto, Venezia
  - Department of Neurology, Sant'Andrea Hospital, Vercelli
  - Department of Neurology and Stroke Unit, Arzignano Azienda ULSS 8 Berica, Vicenza
  - Department of Neurology and Stroke Unit, San Bortolo Hospital, Vicenza
  - Stroke Unit, ASST Vimercate, Vimercate
  - Department of Neurology and Stroke Unit, Guzzardi Hospital, Vittoria

REFERENCES:
- [Background] Wang Y, Wang Y, Zhao X, Liu L, Wang D, Wang C, Wang C, Li H, Meng X, Cui L, Jia J, Dong Q, Xu A, Zeng J, Li Y, Wang Z, Xia H, Johnston SC; CHANCE Investigators. Clopidogrel with aspirin in acute minor stroke or transient ischemic attack. N Engl J Med. 2013 Jul 4;369(1):11-9. doi: 10.1056/NEJMoa1215340. Epub 2013 Jun 26. PMID 23803136
- [Background] Kennedy J, Hill MD, Ryckborst KJ, Eliasziw M, Demchuk AM, Buchan AM; FASTER Investigators. Fast assessment of stroke and transient ischaemic attack to prevent early recurrence (FASTER): a randomised controlled pilot trial. Lancet Neurol. 2007 Nov;6(11):961-9. doi: 10.1016/S1474-4422(07)70250-8. Epub 2007 Oct 10. PMID 17931979
- [Background] Johnston SC, Easton JD, Farrant M, Barsan W, Conwit RA, Elm JJ, Kim AS, Lindblad AS, Palesch YY; Clinical Research Collaboration, Neurological Emergencies Treatment Trials Network, and the POINT Investigators. Clopidogrel and Aspirin in Acute Ischemic Stroke and High-Risk TIA. N Engl J Med. 2018 Jul 19;379(3):215-225. doi: 10.1056/NEJMoa1800410. Epub 2018 May 16. PMID 29766750
- [Background] Johnston SC, Amarenco P, Denison H, Evans SR, Himmelmann A, James S, Knutsson M, Ladenvall P, Molina CA, Wang Y; THALES Investigators. Ticagrelor and Aspirin or Aspirin Alone in Acute Ischemic Stroke or TIA. N Engl J Med. 2020 Jul 16;383(3):207-217. doi: 10.1056/NEJMoa1916870. PMID 32668111
- [Derived] De Santis F, Ornello R, De Matteis E, D'Anna L, Romoli M, Tassinari T, Saia V, Cenciarelli S, Bedetti C, Padiglioni C, Censori B, Puglisi V, Vinciguerra L, Guarino M, Barone V, Zedde M, Grisendi I, Diomedi M, Bagnato MR, Petruzzellis M, Mezzapesa DM, Inchingolo V, Cappellari M, Zivelonghi C, Candelaresi P, Andreone V, Rinaldi G, Bavaro A, Cavallini A, Piscaglia MG, Terruso V, Mannino M, Pezzini A, Frisullo G, Muscia F, Paciaroni M, Mosconi MG, Zini A, Leone R, Palmieri C, Cupini LM, Marcon M, Tassi R, Sanzaro E, Papiri G, Viticchi G, Orsucci D, Falcou A, Beretta S, Tarletti R, Nencini P, Rota E, Sepe FN, Ferrandi D, Caputi L, Volpi G, La Spada S, Beccia M, Rinaldi C, Mastrangelo V, Di Blasio F, Invernizzi P, Pelliccioni G, De Angelis MV, Bonanni L, Ruzza G, Caggia EA, Russo M, Tonon A, Acciarri MC, Anticoli S, Roberti C, Scaglione G, Pistoia F, Fortini A, De Boni A, Sanna A, Chiti A, Barbarini L, Caggiula M, Masato M, Del Sette M, Passarelli F, Bongioanni MR, De Michele M, Ricci S, Sacco S, Foschi M. Real-world outcomes following dual antiplatelet therapy in mild-to-moderate ischemic stroke with anterior versus posterior circulation infarct: a READAPT study propensity matched analysis. Ther Adv Neurol Disord. 2025 Jul 12;18:17562864251351100. doi: 10.1177/17562864251351100. eCollection 2025. PMID 40661752
- [Derived] De Matteis E, De Santis F, Foschi M, Romoli M, Tassinari T, Saia V, Cenciarelli S, Bedetti C, Padiglioni C, Censori B, Puglisi V, Vinciguerra L, Guarino M, Barone V, Zedde M, Grisendi I, Maestrini I, Bagnato MR, Petruzzellis M, Mezzapesa DM, Di Viesti P, Inchingolo V, Cappellari M, Zenorini M, Candelaresi P, Andreone V, Rinaldi G, Bavaro A, Cavallini A, Moraru S, Piscaglia MG, Terruso V, Mannino M, Pezzini A, Frisullo G, Muscia F, Paciaroni M, Mosconi MG, Zini A, Leone R, Palmieri C, Cupini LM, Marcon M, Tassi R, Sanzaro E, Paci C, Viticchi G, Orsucci D, Falcou A, Diamanti S, Tarletti R, Nencini P, Rota E, Sepe FN, Ferrandi D, Caputi L, Volpi G, La Spada S, Beccia M, Rinaldi C, Mastrangelo V, Di Blasio F, Invernizzi P, Pelliccioni G, De Angelis MV, Bonanni L, Ruzza G, Caggia EA, Russo M, Tonon A, Acciarri MC, Anticoli S, Roberti C, Manobianca G, Scaglione G, Pistoia F, Fortini A, De Boni A, Sanna A, Chiti A, Barbarini L, Caggiula M, Masato M, Del Sette M, Passarelli F, Bongioanni MR, Toni D, Ricci S, Sacco S, Ornello R; READAPT Study Group. Real-World Dual Antiplatelet Therapy Use Exceeds Randomized Trials Boundaries With Possible Safety Issues in Patients With Large Artery Atherosclerosis-Insights From the READAPT Study. Eur J Neurol. 2025 Apr;32(4):e70163. doi: 10.1111/ene.70163. PMID 40265654
- [Derived] Foschi M, D'Anna L, De Matteis E, De Santis F, Romoli M, Tassinari T, Saia V, Cenciarelli S, Bedetti C, Padiglioni C, Censori B, Puglisi V, Vinciguerra L, Guarino M, Barone V, Zedde M, Grisendi I, Diomedi M, Bagnato MR, Petruzzellis M, Mezzapesa DM, Di Viesti P, Inchingolo V, Cappellari M, Zivelonghi C, Candelaresi P, Andreone V, Rinaldi G, Bavaro A, Cavallini A, Moraru S, Piscaglia MG, Terruso V, Mannino M, Pezzini A, Frisullo G, Muscia F, Paciaroni M, Mosconi MG, Zini A, Leone R, Palmieri C, Cupini LM, Marcon M, Tassi R, Sanzaro E, Papiri G, Paci C, Viticchi G, Orsucci D, Falcou A, Beretta S, Tarletti R, Nencini P, Rota E, Sepe FN, Ferrandi D, Caputi L, Volpi G, La Spada S, Beccia M, Rinaldi C, Mastrangelo V, Di Blasio F, Invernizzi P, Pelliccioni G, De Angelis MV, Bonanni L, Ruzza G, Caggia EA, Russo M, Tonon A, Acciarri MC, Anticoli S, Roberti C, Manobianca G, Scaglione G, Pistoia F, Fortini A, De Boni A, Sanna A, Chiti A, Barbarini L, Caggiula M, Masato M, Del Sette M, Passarelli F, Bongioanni MR, De Michele M, Ricci S, Ornello R, Sacco S; READAPT Study Group. Exploring Sex Differences in Outcomes of Dual Antiplatelet Therapy for Patients With Noncardioembolic Mild-to-Moderate Ischemic Stroke or High-Risk Transient Ischemic Attack: A Propensity-Matched Analysis of the READAPT Study Cohort. Stroke. 2025 Feb;56(2):305-317. doi: 10.1161/STROKEAHA.124.049210. Epub 2024 Dec 9. PMID 39648888
- [Derived] Ornello R, Foschi M, De Santis F, Romoli M, Tassinari T, Saia V, Cenciarelli S, Bedetti C, Padiglioni C, Censori B, Puglisi V, Vinciguerra L, Guarino M, Barone V, Zedde M, Grisendi I, Diomedi M, Bagnato MR, Petruzzellis M, Mezzapesa DM, Di Viesti P, Inchingolo V, Cappellari M, Zivelonghi C, Candelaresi P, Andreone V, Rinaldi G, Bavaro A, Cavallini A, Moraru S, Querzani P, Terruso V, Mannino M, Pezzini A, Frisullo G, Muscia F, Paciaroni M, Mosconi MG, Zini A, Leone R, Palmieri C, Cupini LM, Marcon M, Tassi R, Sanzaro E, Paci C, Viticchi G, Orsucci D, Falcou A, Beretta S, Tarletti R, Nencini P, Rota E, Sepe FN, Ferrandi D, Caputi L, Volpi G, La Spada S, Beccia M, Rinaldi C, Mastrangelo V, Di Blasio F, Invernizzi P, Pelliccioni G, De Angelis MV, Bonanni L, Ruzza G, Caggia EA, Russo M, Tonon A, Acciarri MC, Anticoli S, Roberti C, Manobianca G, Scaglione G, Pistoia F, Fortini A, De Boni A, Sanna A, Chiti A, Barbarini L, Caggiula M, Masato M, Del Sette M, Passarelli F, Bongioanni MR, Toni D, Ricci S, De Matteis E, Sacco S; READAPT Study Group. Combining Intravenous Thrombolysis and Dual Antiplatelet Treatment in Patients With Minor Ischemic Stroke: A Propensity Matched Analysis of the READAPT Study Cohort. J Am Heart Assoc. 2024 Aug 20;13(16):e036275. doi: 10.1161/JAHA.124.036275. Epub 2024 Aug 9. PMID 39119964
- [Derived] De Matteis E, De Santis F, Ornello R, Censori B, Puglisi V, Vinciguerra L, Giossi A, Di Viesti P, Inchingolo V, Fratta GM, Diomedi M, Bagnato MR, Cenciarelli S, Bedetti C, Padiglioni C, Tassinari T, Saia V, Russo A, Petruzzellis M, Mezzapesa DM, Caccamo M, Rinaldi G, Bavaro A, Paciaroni M, Mosconi MG, Foschi M, Querzani P, Muscia F, Gallo Cassarino S, Candelaresi P, De Mase A, Guarino M, Cupini LM, Sanzaro E, Zini A, La Spada S, Palmieri C, Sepe FN, Beretta S, Paci C, Caggia EA, De Angelis MV, Bonanni L, Volpi G, Tassi R, Pistoia F, Scoditti U, Tonon A, Viticchi G, Ruzza G, Nencini P, Cavallini A, Toni D, Ricci S, Sacco S; READAPT Study Group. Divergence Between Clinical Trial Evidence and Actual Practice in Use of Dual Antiplatelet Therapy After Transient Ischemic Attack and Minor Stroke. Stroke. 2023 May;54(5):1172-1181. doi: 10.1161/STROKEAHA.122.041660. Epub 2023 Mar 23. PMID 36951052

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT05476081/Prot_SAP_000.pdf